CLINICAL TRIAL: NCT00090558
Title: Effect of Nitric Oxide Donor on Endothelial Progenitor Cells in Patients With Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040268; 04-H-0268
Record Dates: First submitted 2004-08-27; First posted 2004-08-27 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-09

CONDITIONS: Coronary Artery Disease
Keywords: Atherosclerosis; Bone Marrow; Exercise; Endothelium; Nitroglycerin; Coronary Artery Disease; CAD
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Motor Activity | interventions — Nitroglycerin

INTERVENTIONS:
Drug: nitroglycerin

SUMMARY:
Regular exercise reduces the risk of heart problems, in part because it improves the work of the endothelium (the cells that line blood vessels). Exercise appears to release precursor cells from the bone marrow that will later become endothelial cells. A molecule called nitric oxide (NO) appears to be involved in this release. However, some heart patients do not improve their endothelial function despite regular exercise. The researchers believe that the heart disease in these patients may interfere with the normal relationship between exercise and endothelial function. This study is designed to test whether giving a patient nitroglycerin (which is converted to NO in the bloodstream) will increase the release of endothelial precursor cells from the bone marrow. If the study succeeds, it may lead to improved healing of arteries in heart disease patients.

Adults may be eligible for this study if they have coronary artery disease and do not take nitroglycerin or nitroglycerin-like medication on a daily basis.

Volunteers will be admitted to the Clinical Center on 2 separate nights at least 1 week apart. On the morning after each admission, volunteers will have blood drawn from an arm vein for laboratory tests, and then walk on a treadmill until fatigue or discomfort prevents further exercise, or until asked to stop. On one of their admissions, volunteers will receive 1 tablet of nitroglycerin under the tongue shortly before the treadmill test. Volunteers will be monitored by EKGs and blood pressure tests during the treadmill tests, and will have more blood drawn at about 15 minutes and 24 hours after each treadmill test. Researchers will examine the levels of endothelial precursor cells and nitric oxide in the blood samples taken before and after exercise.

DETAILED DESCRIPTION:
Exercise training has long been recommended as a means of improving cardiac function and reducing morbidity and mortality in patients with coronary artery disease (CAD). One mechanism of benefit may be through improved endothelial function and enhanced nitric oxide (NO) bioactivity, which may improve blood flow to exercising skeletal muscle and to the myocardium. We have recently determined in a collaborative study with the Suburban Hospital, however, that many CAD patients do not show improved endothelial function despite compliant participation in a three month cardiac rehabilitation program with exercise three times weekly. The initial data from this study suggest that improvement in endothelial function may be dependent on the release of endothelial progenitor cells (EPCs) from the bone marrow into the circulation in response to the stimulus of repetitive exercise, with the potential of repairing damaged endothelium and improving endothelial function and NO release. Thus, patients who have poor EPC mobilization responses to exercise may have limited capacity to improve endothelial function over time and, conversely, patients with higher EPC mobilization responses to exercise may show improved endothelial function as a result of vascular repair. Animal models indicate that NO is necessary for EPC mobilization during exercise, likely through nitrosation reactions with key signaling proteins within bone marrow. In many CAD patients, NO release from endothelium and transport in blood to bone marrow may be compromised because of atherosclerotic vascular disease, and thus limit EPC mobilization and vascular repair. We hypothesize that the exogenous administration of NO to CAD patients may enhance EPC mobilization from bone marrow in response to exercise. If successful, administration of an NO donor (such as nitroglycerin) prior to exercise may extend the benefit of exercise to endothelial function-and thus cardiovascular risk-in a larger segment of CAD patients participating in cardiac rehabilitation programs.

ELIGIBILITY:
PATIENT INCLUSION CRITERIA

1. Adults older than 21 years.
2. Coronary artery disease established by angiography.
3. No myocardial infarction within 1 month.
4. Left ventricular ejection fraction greater than 30%.
5. No congestive heart failure symptoms within 2 months.
6. No associated medical, neurological or orthopedic condition that might prohibit safe performance of exercise.
7. Subject understands protocol and provides written, informed consent in addition to willingness to comply with specified follow-up evaluations.

PATIENT EXCLUSION CRITERIA

1. Significant structural heart disease (e.g. hypertrophic or dilated cardiomyopathy, valvular heart disease) as determined by echocardiography.
2. History of recent (within 2 months) rest or nocturnal angina
3. Organic nitrate (e.g., nitroglycerin) use other than study medication within 24 hours of exercise testing
4. Hypersensitivity to organic nitrates.
5. Women of childbearing age unless recent pregnancy test is negative.
6. Lactating women.

ELIGIBILITY CRITERIA - HEALTHY SUBJECTS

Healthy subjects must be older than 50 years of age (to approximate the anticipated age of CAD patients), without known CAD, and be free of the following risk factors: blood pressure greater than 140/90 mmHg, fasting glucose greater than 110 mg/dL, smoking, total cholesterol greater than 250 mg/dL. Healthy subjects taking chronic prescription medications will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-08; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States